CLINICAL TRIAL: NCT00291889
Title: Evaluate the Safety, Reactogenicity & Immunogenicity of 2 Antigen Dose Levels of GSK Biologicals' Candidate Tuberculosis Vaccine, Mtb72F/AS02 to Healthy PPD-negative Volunteers Aged 18 to 45 Yrs
Brief Title: Safety and Immunogenicity of GSK Biological's Candidate Tuberculosis Vaccine Mtb72F/AS02 in Healthy PPD-negative Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 102039
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Tuberculosis (TB)
MeSH Terms: conditions — Tuberculosis

INTERVENTIONS:
Biological: Mtb72F/AS02.

SUMMARY:
Vaccination against tuberculosis (TB) /healthy PPD-negative adults aged 18 to 45 years.Three doses of primary vaccination followed by a booster dose after completion of primary vaccination course. Booster vaccination will be given only to subjects receiving the candidate tuberculosis vaccines and not to the subjects receiving active comparators or control.

DETAILED DESCRIPTION:
The safety and immunogenicity of 2 antigen doses in PPD-negative adults will be evaluated. In addition, 2 active comparator groups of volunteers will receive the vaccine alone without an immunostimulant and 1 control group will receive the adjuvant (AS02) alone to assess the true effect of the candidate tuberculosis vaccine (Mtb72F/AS02).

ELIGIBILITY:
INCLUSION CRITERIA:

* Written informed consent
* Healthy PPD-negative volunteers aged 18 to 45 years
* No evidence of pulmonary pathology (i.e. acute or chronic pulmonary disease; past TB infection/disease) as confirmed by chest X-ray.
* Seronegative for HIV 1 and 2, HBsAg, and HCV
* Clinically normal laboratory values for creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, complete blood count (CBC) and differential, haemoglobin, platelet count and urinalysis.
* Females : Non pregnant, must use adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

EXCLUSION CRITERIA:

* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* History of prior Bacillus Calmette-Guérin (BCG) vaccination.
* History of documented exposure to Mycobacterium tuberculosis
* History of prior vaccination with experimental Mycobacterium Tuberculosis vaccines or experimental products containing MPL or QS21.
* Any confirmed or suspected immunosuppressive or immunodeficient condition; or family history of congenital or hereditary immunodeficiency.
* History of hypersensitivity to vaccines or vaccine components
* History of any acute or chronic illness or medication that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2004-07; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited symptoms during the 7-day follow-up period, unsolicited symptoms during the 30-day follow-up period, grade 3 vaccine related local and general symptoms during the 30-day follow-up and serious adverse events during the entire study

SECONDARY OUTCOMES:
Immunogenicity as assessed by humoral and CMI response.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium